CLINICAL TRIAL: NCT04896060
Title: The Impact of the Food Environment and Psychosocial Stress From the COVID-19 Pandemic on Eating Behavior and Weight Change
Brief Title: The Impact of the COVID-19 Pandemic on Eating Behavior and Weight Change
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000172; 000172-DK
Record Dates: First submitted 2021-05-19; First posted 2021-05-21 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12-23

CONDITIONS: COVID-19; Obesity
Keywords: Obesity; Food Intake; Food Insecurity; Resilience; Unpredictability; Natural History
MeSH Terms: conditions — COVID-19; Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ecological Momentary Assessment (EMA) volunteers: Volunteers with access to mobile device with Wi-Fi and data recruited for an additional 1-week daily assessment study utilizing EMA to examine COVID-19 related stress and eating behavior in real-time
- General global population volunteers: Newly recruited volunteers 18 and above from the general global population that agree to participate in the COVID study
- NIDDK-Phoenix study volunteers: Previous research participants, who signed consents that allow data sharing that agree to participate in the COVID study

SUMMARY:
Background:

The indirect effects of the COVID-19 pandemic on mental health are of increasing concern. Perceived stress can lead to binge eating and weight gain. Researchers want to learn more about the relationship between eating behavior and the pandemic.

Objective:

To study how the stress of the COVID-19 pandemic is affecting eating behaviors and weight.

Eligibility:

English-speaking adults ages 18 and older who have access to a computer or smartphone connected to the internet.

Design:

This is an online study. Participants will answer surveys through the study website.

Participants will complete a one-time survey. It will ask about their experiences throughout the COVID-19 pandemic, their socioeconomic standing, their mental and physical health, and their eating habits. They will have the option to repeat the survey once a month for the next 12 months. This will show changes in their thoughts and behaviors over time. They will provide their email address to get survey links.

Participants will also have the option to complete a 2-minute survey on their smartphone. They will complete the survey daily for 7 days in a row. It will ask about their stress and eating behavior in real time, in their home environment. They will provide their phone number to get survey links via text message.

If a participant has taken part in a previous NIH study on the Phoenix AZ campus, they will be asked to share their first and last name, date of birth, and email address. This information will be used to connect data from this study to their past data.

Participation is typically 25 minutes but may last up to 1 year.

***To participate in this study go to the REDCap study link: https://redcap.link/nihcovidstudy.***...

DETAILED DESCRIPTION:
Study Description:

We will recruit previous NIDDK study participants as well as newly recruited individuals from the general population to examine how the COVID-19 pandemic has exacerbated the impact of psychosocial stressors that impact eating behavior and weight. The study will describe the relationship between specific COVID-19 related stressors (e.g. fear of becoming sick) and self-rated measures of food insecurity, unpredictability, perceived stress, behavioral health dysfunction, eating behaviors and weight change among a range of participants including previous NIDDK-Phoenix study volunteers and various newly recruited volunteers from the general global population. Participants will be invited to enroll in a follow- up study which will involve completing additional surveys on a monthly basis for 12 months. A smaller U.S. only cohort of these participants may also enroll in a 2 minute daily at-home survey study for 1-weekthat will utilize Ecological Momentary Assessment (EMA) to examine stress and eating behavior in real-time, in the home environment. Participants will complete an online consent form and online survey through a secure weblink (REDCap). Because the situation with the COVID-19 pandemic is rapidly changing, survey data collection is an effective way to measure outcomes at multiple time points with relatively low subject burden.

Objectives:

Primary Objective: to examine the food environment and psychosocial stressors related to COVID-19 with self-reported measures of behavioral health symptoms, eating behaviors and weight.

Secondary Objective: to determine whether sociodemographic, existing behavioral health dysfunction, or environmental condition moderates this relationship and to identify risk and resilience factors among study participants regarding the impact of the COVID-19 pandemic on eating behavior and weight.

Endpoints:

Primary Endpoints: measures of eating behavior and body weight. These endpoints will be measured repeatedly using an online platform (REDCap) at baseline and then monthly for up to 12 months. We also plan to examine these COVID-19 related measures with previously collected phenotypic data (e.g. biological samples and behavioral data) from former NIDDK-Phoenix participants.

Secondary Endpoints: in addition to those outlined as primary endpoints, we will examine data gathered from demographic forms and additional questionnaires measuring environmental conditions and psychosocial stress.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all the following criteria:

1. 18 years of age or older
2. Able to read and write English
3. Consistent access to computer or mobile devices connected to the internet
4. Able to provide informed consent online and/or in-person

In order to be eligible to participate in the EMA arm of the study, an individual must meet all the following criteria:

1. Access to a mobile device with WI-FI and data

EXCLUSION CRITERIA:

1. Non-English-speaking individuals.

Non-English-speaking subjects as a population will be excluded from participation in this protocol. The primary aim of the protocol relates to the questionnaires administered to the participants online. There are currently no validated, translated forms of these questionnaires available; therefore, we will restrict enrollment to English speaking subjects only.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers of any health status, sex, or gender who are at least 18 years old. English-speaking. Previously consented NIDDK Phoenix study volunteers and new participants from the general population. Conducted online so physical location is unrestricted.
Sampling Method: Non-Probability Sample
Enrollment: 5056 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Nighttime Eating Behavior | Baseline and 12 months
  2 questions taken from the Night Eating Diagnostic Questionnaire (NEDQ), a self-report questionnaire containing 14 questions about eating after the evening meal and waking up in the night to eat. Symptoms are rated on a 5-point Likert-type scale, which are then summed to obtain a NEQ Global Score.
The Intuitive Eating Scale-2 (IES-2) | Baseline and 12 months
  The IES-2 consists of 23-items measuring individuals tendency to follow their physical hunger and satiety cues when determining when, what, and how much to eat. Scores are rated on a 5-point Likert scale ranging from strongly disagree to strongly agree. Items are summed and an average score is computed for the entire scale and its four subscales.
Three Factor Eating Questionnaire (TFEQ) | Baseline and 12 months
  TFEQ consists of 18 items on a 4-point response scale (definitely true/mostly true/mostly false/definitely false) (scores recorded on a 0-100 scale). Higher scores in the respective scales are indicative of greater cognitive restraint, uncontrolled, or emotional eating.
Loss of Control Eating | Baseline and 12 months
  2 questions to assess eating a large amount of food and sense of loss of control over one s eating behavior
Food Frequency Questionnaire (FFQ) | Baseline and 12 months
  Semiquantitative self-administered questionnaire that estimates average daily intake of foods, drinks, energy, and major nutrients out of about 124 different foods.
Changes in self-reported weight | Baseline and 12 months
  Changes in self-reported weight from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marci E Gluck, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Willig M, Cabeza de Baca T, J Stinson E, M Trevino-Alvarez A, Rodzevik T, B Votruba S, C Lameman C, Krakoff J, Gluck ME. The impact of COVID-19 fear during the later stages of the pandemic on maladaptive eating, psychological distress and body weight: a global cross-sectional study. BMC Public Health. 2025 Apr 11;25(1):1365. doi: 10.1186/s12889-025-22444-6. PMID 40217216
- See also: https://redcap.link/nihcovidstudy — https://redcap.link/nihcovidstudy